CLINICAL TRIAL: NCT05719545
Title: A Longitudinal Cohort of Patients With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention
Brief Title: A Cohort of Patients Undergoing Percutaneous Coronary Intervention
Acronym: APCIcohort
Status: Recruiting | Type: Observational
Sponsor: Su Guohai (Other)
Collaborators: Shandong First Medical University (Other)
Responsible Party: Sponsor-Investigator, Su Guohai, Professor, Jinan Central Hospital
Organization: Jinan Central Hospital (Other)
Other Study IDs: 2021-206-02
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention; Myocardial Infarction; Unstable Angina
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and fecal samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the risk factors involved in the occurrence and prognosis of the patients with acute coronary syndrome, patients undergoing percutaneous coronary intervention will be recruited and followed up for at least 2 years.

DETAILED DESCRIPTION:
Patients with acute coronary syndrome undergoing percutaneous coronary intervention will be recruited and prospectively followed up for the incidence of major adverse cardiovascular events (MACE events), including all-cause mortality, cardiovascular mortality, ischemic stroke. Blood and fecal samples will be collected for further analysis. The basic and clinical information will be collected such as diagnosis, medical history, laboratory test results, therapy methods, prognosis and follow-up information. The risk factors involved in the occurrence and prognosis of acute coronary syndrome will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as acute coronary syndrome and needed to undergo percutaneous coronary intervention.
* >18 years old.

Exclusion Criteria:

* With malignant tumors, acute infectious diseases and advanced liver diseases.
* Won't sign an inform consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome undergoing percutaneous coronary intervention.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | 2-year outcome and long-term outcome
  all-cause mortality, cardiovascular mortality, ischemic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Guohao Su, doctor, Principal Investigator — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China